CLINICAL TRIAL: NCT03579667
Title: Lipid Profile and Weight After Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Responsible Party: Principal Investigator, Hilde Kristin Brekke, Professor, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017/450
Record Dates: First submitted 2018-06-25; First posted 2018-07-06 (Actual); Last update posted 2021-10-27 (Actual); Status verified 2021-10

CONDITIONS: Cardiovascular Risk Factor; Body Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diet intervention (Experimental)
  Interventions: Behavioral: Diet intervention
- Control (No Intervention)

INTERVENTIONS:
Behavioral: Diet intervention — 12-week program of dietary behavior modification treatment (LEVA-method by Bertz et al, Am J Clin Nutr 2012;96:698.), leading to 6 kg weight loss (0.5 kg per week) and a healthier diet (less sugar, snacks, full fat products, more vegetables and fruit, smaller portion sizes). Weight is monitored by phone contact every second week. After 12 weeks, the women are followed up by e-mail contact for 9 additional months.
  Arms: Diet intervention

SUMMARY:
A randomized controlled trial aiming to investigate the effects of diet behavior intervention postpartum on body weight and lipid and metabolite profile in overweight and obese women in Oslo, Norway

ELIGIBILITY:
Inclusion Criteria:

* Women admitted to Adipol, Oslo University Hospital, Norway (outpatient clinic for women with overweight or obesity during pregnancy)

Exclusion Criteria:

* Twin birth,
* Non-Norwegian speaking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women With prepregnant overweight or obesity (BMI>27)
Enrollment: 30 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Changes in body weight (kg) between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured in light clothing without shoes. Together with measured height (m) will be used to calculate Body Mass Index.
Changes in markers of lipid- and glucose metabolism between visits | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured in mmol/l: total cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides and glucose In percentage: HbA1c In pmol/l: insulin.

SECONDARY OUTCOMES:
Changes in lipid subclasses (mmol/l), lipoprotein size (nm) and apolipoproteins between visits | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  In g/l: apolipoprotein (apo) B and apo A1. In mmol/l: lipoprotein (a)
Changes in blood pressure, diastolic and systolic between visits | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured after 5 min rest, mean of 2 measurements (mmHg)
Changes in waist and hip (cm) circumference between visits | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  A measuring tape specifically designed for waist circumference (Seca) will be used according to a standardized procedure Measurements will be taken against the skin at the approximate midpoint between the lower margin of the last palpable rib and the top of the iliac crest. Hip is measured over the widest point on the buttocks
Changes in body composition (fat free mass in kg and fat mass in kg) between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured by Bioelectrical impedance
Changes in circulating inflammation markers such as cytokines, high sensitivity C-Reactive Protein, C-Reactive Protein (CRP) and microCRP between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured in mg/l
Changes in plasma metabolomics such as lactate, pyruvate, citrate and amino acids between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured in mmol/l
Changes in PBMC (peripheral blood mononuclear cell) gene expression levels of markers of inflammation and lipid metabolism between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Changes in levels of markers of inflammation and lipid metabolism at PBMC gene expression level.
Changes in hemostatic markers such as plasminogen activator inhibitor-1 (PAI-1) antigen and von Willebrand factor (vWF) between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  PAI-1 measured in ng/mL, vWF measured in IU/dl
Changes in hormones such as prolactin, estradiol, progesterone between visits | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured in nmol/l
Changes in markers of micronutrient status such as Hb and vitamin D between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Measured in g/dl (Hb), nm/l (vit D)
Changes in dietary intake and Food Choice by food frequency questionnaire at each of the 3 visits | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Energy (KJ/kcal), macronutrients and micronutrients will be calculated in Norwegian Food database program. The diet questionnaire is optically readable and has 11-pages. It contains 180 food items grouped by food groups; breads, spreads, cereals, milk, yoghurt, drinks (cold, warm, alcoholic), dinner foods (potatoes, rice, pasta, vegetables), sauces and dressings, fats, fruits, desserts/cakes/sweets/snacks, diet supplements. Frequencies are most often given in 9 categories, varying from rarely/never to 4 or more times per day, depending on food category. Portion-sizes are given as typical household units: slices, glasses, cups, pieces, spoons and ladle.
Changes in physical activity between visits. | Visit 1 (8 weeks postpartum, visit 2 (6 months postpartum) and visit 3 (15 months postpartum)]
  Questions are asked about physical activity before and during pregnancy as well as current postpartum visit. At these timepoints, four dimensions of activities are examined; 1) everyday activities (four response categories from inactive (0 points) to heavy physical work (3 points)), 2) transportation (two response categories: passive (car/public transport, 0p), active (walk or bike 1p)), 3) leisure time/outdoor activity (five response categories from rarely (0p) to 4 times/week or more (4p)) and 4) 30 min continuous physical activity with increased pulse/being short-winded (five response categories from rarely (0p) to 4 times/week or more (4p)). Participants receive a score for each of the four dimensions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oslo, Oslo, Norway

REFERENCES:
- [Derived] Ohman EA, Fossli M, Ottestad I, Holven KB, Ulven SM, Loland BF, Brekke HK. Dietary treatment postpartum in women with obesity reduces weight and prevents weight gain: a randomised controlled trial. BMC Pregnancy Childbirth. 2023 Sep 26;23(1):695. doi: 10.1186/s12884-023-05976-w. PMID 37752466